CLINICAL TRIAL: NCT04090528
Title: Phase II Trial of pTVG-HP DNA Vaccine With or Without pTVG-AR DNA Vaccine and Pembrolizumab in Patients With Castration-Resistant, Metastatic Prostate Cancer
Brief Title: pTVG-HP DNA Vaccine With or Without pTVG-AR DNA Vaccine and Pembrolizumab in Patients With Castration-Resistant, Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Madison Vaccines Incorporated (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW18037; 2018-0938 (Other: Institutional Review Board); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); A534260 (Other: UW Madison); NCI-2019-07273 (Registry Identifier: NCI Trial ID); Protocol Version 2/10/2025 (Other: UW Madison)
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Castration-resistant Prostate Cancer; Metastatic Cancer; Prostate Cancer
Keywords: immunotherapy; prostate cancer; vaccine; DNA vaccine; pTVG-HP; pTVG-AR; androgen receptor; prostatic acid phosphatase; pembrolizumab
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms; Bulbo-Spinal Atrophy, X-Linked | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 1:1 randomized, open-label, multi-institution phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: One DNA vaccine (Experimental): 100 µg pTVG-HP administered intradermally (i.d.) days 1, 8 plus 200 mg Pembrolizumab, administered intravenously on day 1 of 21-day cycles (for 8 cycles)
  Following cycle 8, subsequent 21-days cycles: Pembrolizumab 200 mg IV day 1 of 21-day cycles
  In the event of PSA rise (25% increase over cycle 9 day 1, minimum of 2 ng/ml), and no evidence of radiographic progression, participants will receive 4 additional vaccine booster cycles: 100 µg pTVG-HP i.d. days 1, 8 + 200 mg pembrolizumab IV day 1 of 21-day cycles x 4 cycles
  Interventions: Biological: pTVG-HP; Drug: Pembrolizumab
- Arm 2: Two DNA vaccines (Experimental): 100 µg pTVG-AR administered intradermally (i.d.) on days 1, 8 plus 200 mg Pembrolizumab administered intravenously day 1 of 21-day cycles, for cycles 1, 2, 5, and 6 alternating with 100 µg pTVG-HP administered intradermally (i.d.) on days 1, 8 plus 200 mg Pembrolizumab administered intravenously day 1 of 21-day cycles, for cycles 3, 4, 7, and 8.
  Following cycle 8, subsequent 21-days cycles: Pembrolizumab 200 mg IV day 1 of 21-day cycles
  In the event of PSA rise (25% increase over cycle 9 day 1, minimum of 2 ng/ml), and no evidence of radiographic progression, participants will receive 4 additional vaccine booster cycles: 100 µg pTVG-AR i.d days 1, 8 + 200 mg pembrolizumab IV day 1 of q 21-day cycles, for cycles 1 and 2 followed by 100 µg pTVG-HP i.d. days 1, 8 + 200 mg pembrolizumab IV day 1 in 21-day cycles, for cycles 3 and 4
  Interventions: Biological: pTVG-HP; Biological: pTVG-AR; Drug: Pembrolizumab

INTERVENTIONS:
Biological: pTVG-HP — pTVG-HP is a plasmid DNA, produced in E. coli, that encodes the complementary deoxyribonucleic acid (cDNA) for human prostatic acid phosphatase (PAP).
Biological: pTVG-AR — pTVG-AR is a plasmid DNA
  Arms: Arm 2: Two DNA vaccines
Drug: Pembrolizumab — Pembrolizumab is a human programmed death receptor-1 (PD-1)-blocking antibody indicated for the treatment of patients with multiple different types of cancer.
  Other Names: Keytruda

SUMMARY:
This trial will evaluate the use of one versus two DNA vaccines, delivered concurrently with PD-1 blockade using pembrolizumab followed by treatment with pembrolizumab alone, and delivered over a prolonged period of time (for a maximum of 2 years (32 cycles) or until radiographic progression) on the treatment of castrate-resistant, metastatic prostate cancer. The hypothesis to be tested is that delivering two vaccines with PD-1 blockade will elicit a greater frequency and magnitude of tumor-directed CD8+ T cells, and thereby increase the percentage of patients experiencing objective anti-tumor effect as measured by PSA declines and/or objective radiographic responses. Participants must be 18 years of age or older and can expect to be on treatment for 2 years (32 cycles) and on study for up to 7 years (including 5 years of follow up via phone).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate)
* Metastatic disease as evidenced by the presence of soft tissue and/or bone metastases on imaging studies (CT of abdomen/pelvis, bone scintigraphy)
* Castrate-resistant disease, defined as follows:

  * All participants must have received (and be receiving) standard of care androgen deprivation treatment (surgical castration versus GnRH analogue or antagonist treatment); subjects receiving Gonadotropin-releasing hormone (GnRH) analogue or antagonist must continue this treatment throughout the time on this study.
  * Participants may or may not have been treated previously with a nonsteroidal antiandrogen. For participants previously treated with an antiandrogen, they must be off use of anti-androgen for at least 28 days before day 1 (for flutamide, apalutamide, enzalutamide, or other 2nd generation AR antagonists) or 6 weeks (for bicalutamide or nilutamide) prior to registration. Moreover, participants who demonstrate an anti-androgen withdrawal response, defined as a > 25% decline in PSA within 4-6 week of stopping a nonsteroidal antiandrogen, are not eligible until the PSA rises above the nadir observed after antiandrogen withdrawal.
  * Participants must have a castrate serum level of testosterone (< 50 ng/dL) within 6 weeks of day 1
* Progressive disease while receiving androgen deprivation therapy defined by any one of the following as per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) bone scan criteria or RECIST 1.1 during or after completing last therapy:

  * PSA: At least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, with the final value > 2.0 ng/mL.
  * Measurable disease: > 50% increase in the sum of the cross products of all measurable lesions or the development of new measurable lesions. The short axis of a target lymph node must be at least 15 mm by spiral CT to be considered a target lesion
  * Non-measurable (bone) disease: The appearance of two or more new areas of uptake on bone scan (or Sodium Fluoride (NaF) positron emission tomography-computed tomography (PET/CT)) consistent with metastatic disease compared to previous imaging during castration therapy. The increased uptake of pre-existing lesions on bone scan will not be taken to constitute progression, and ambiguous results must be confirmed by other imaging modalities (e.g. X-ray, CT or MRI).
* Prior treatment with abiraterone or enzalutamide is permitted, but participants must have weaned to a daily corticosteroid dose equivalent of no more than 5 mg prednisone daily for at least 28 days prior to day 1.
* Life expectancy of at least 6 months
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Adequate hematologic, renal, liver, and coagulation function as evidenced by the following within 6 weeks of day 1:

  * White Blood Cells (WBC) >/= 2000 / mm3
  * Absolute Neutrophil Count (ANC) >/= 1500 / mm3
  * Hemoglobin (HgB) >/= 9.0 gm/dL (Participants must not have received a blood transfusion within 14 days)
  * Platelets >/= 100,000 / mm3
  * Creatinine </= 1.5 x institutional upper limit of normal (ULN)
  * Total bilirubin </= 1.5 x institutional ULN OR direct bilirubin </= ULN for participants with total bilirubin levels > 1.5 x ULN
  * Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) </= 2.5 x institutional upper limit of normal
  * Prothrombin Time (PT) or International Normalized Ratio (INR) </= 1.5 x ULN unless participant is receiving anticoagulant therapy and PT is within therapeutic range of intended use of anticoagulant (only required for participants receiving biopsy)
  * Partial Thromboplastin Time (PTT) </= 1.5 x ULN unless participant is receiving anticoagulant therapy and a PTT is within therapeutic range of intended use of anticoagulant (only required for participants receiving biopsy)
* No known history of human immunodeficiency viruses (HIV 1 and 2), Human T-cell leukemia virus type 1 (HTLV-1), or active Hepatitis B or Hepatitis C
* Participants must be at least 4 weeks from any prior treatments and have recovered (to < Grade 2) from acute toxicity attributed to this prior treatment, unless considered chronic
* A subset of participants (6 participants per treatment arm) treated at the lead University of Wisconsin (UW) site must be willing and able (in the opinion of the treating physician) to undergo two research biopsies for the investigational component of this trial.
* A subset of participants (6 participants per treatment arm) treated at the lead UW site must be willing to undergo NaF PET/CT scans for the investigational component of this trial.
* For those participants who are sexually active, they must be willing to use barrier contraceptive methods, and refrain from donating sperm, during the period of treatment on this trial and for four weeks after the last DNA immunization treatment
* Participants must be informed of the experimental nature of the study and its potential risks, and must sign an Institutional Review Board (IRB)-approved written informed consent form indicating such an understanding

Exclusion Criteria:

* Small cell or other variant (non-adenocarcinoma) prostate cancer histology, unless there is evidence that the tumor expresses PAP
* Participants may not be receiving other investigational agents or be receiving concurrent anticancer therapy other than standard androgen deprivation therapy
* Concurrent bisphosphonate therapy is not excluded, however participants should not start bisphosphonate therapy while on this study; those participants already receiving bisphosphonate therapy should continue at the same dosing and schedule as prior to study entry
* Rapidly progressive symptomatic metastatic disease, as defined by the need for increased opioid analgesics within one month of registration for the treatment of pain attributed to a prostate cancer metastatic lesion; participants receiving opioids must receive approval from the PI for eligibility
* Treatment with any of the following medications within 28 days of day 1, or while on study, is prohibited:

  * Systemic corticosteroids (at doses over the equivalent of 5 mg prednisone daily); inhaled, intranasal or topical corticosteroids are acceptable
  * Prostate Cancer and spes (PC-SPES)
  * Megestrol
  * Ketoconazole
  * 5-α-reductase inhibitors - participants already taking 5-α-reductase inhibitors prior to 28 days prior to registration may stay on these agents throughout the course of therapy, but these should not be started while participants are on study
  * Diethyl stilbesterol
  * Abiraterone
  * Enzalutamide
  * Apalutamide
  * Radium 223 (Xofigo®)
  * Any other hormonal agent or supplement being used with the intent of cancer treatment must be reviewed by the PI for eligibility
* External beam radiation therapy within 4 weeks of registration is prohibited, or anticipated need for radiation therapy (e.g. imminent pathological fracture or spinal cord compression) within 3 months of registration. Participants must have recovered from all radiation-related toxicities and not have had radiation pneumonitis.
* Major surgery within 4 weeks of registration is prohibited
* Prior cytotoxic chemotherapy (for example, but not limited to, docetaxel, mitoxantrone, cabazitaxel) within 28 days of registration is prohibited
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or with any agent directed to another T-cell stimulatory or inhibitory receptor (e.g. CTLA-4, OX-40, CD137).
* Participants with a history of life-threatening autoimmune disease
* Participants with a history of non-infectious pneumonitis that required corticosteroid treatment, or has current pneumonitis
* Participants with a history of allergic reactions to the tetanus vaccine
* Participants who have undergone splenectomy or who have a diagnosis of immunodeficiency
* Participants must not have other active malignancies other than non-melanoma skin cancers or superficial (non-muscle-invasive) carcinoma of the bladder. Participants with a history of other cancers who have been adequately treated and have been recurrence-free for > 3 years are eligible.
* Participants with known brain metastases and/or carcinomatous meningitis
* Participants who have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette - Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Any antibiotic therapy within 1 month of day 1, or anticipated need for antibiotic therapy within 1 month of beginning treatment
* Participants with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Any other medical intervention or condition, which, in the opinion of the PI or treating physician, could compromise participant safety or adherence with the study requirements (including biopsies), or confound results of the study, over the treatment period.
* Any known psychiatric or substance abuse disorders that would interfere with cooperation with the requirement of the trial.
* Participants cannot have concurrent enrollment on other phase I, II, or III investigational treatment studies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2026-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: One DNA Vaccine: 100 µg pTVG-HP administered intradermally (i.d.) days 1, 8 plus 200 mg Pembrolizumab, administered intravenously on day 1 of 21-day cycles (for 8 cycles)
  Following cycle 8, subsequent 21-days cycles: Pembrolizumab 200 mg IV day 1 of 21-day cycles
  In the event of PSA rise (25% increase over cycle 9 day 1, minimum of 2 ng/ml), and no evidence of radiographic progression, participants will receive 4 additional vaccine booster cycles: 100 µg pTVG-HP i.d. days 1, 8 + 200 mg pembrolizumab IV day 1 of 21-day cycles x 4 cycles
  pTVG-HP: pTVG-HP is a plasmid DNA, produced in E. coli, that encodes the complementary deoxyribonucleic acid (cDNA) for human prostatic acid phosphatase (PAP).
  Pembrolizumab: Pembrolizumab is a human programmed death receptor-1 (PD-1)-blocking antibody indicated for the treatment of patients with multiple different types of cancer.
- Arm 2: Two DNA Vaccines: 100 µg pTVG-AR administered intradermally (i.d.) on days 1, 8 plus 200 mg Pembrolizumab administered intravenously day 1 of 21-day cycles, for cycles 1, 2, 5, and 6 alternating with 100 µg pTVG-HP administered intradermally (i.d.) on days 1, 8 plus 200 mg Pembrolizumab administered intravenously day 1 of 21-day cycles, for cycles 3, 4, 7, and 8.
  Following cycle 8, subsequent 21-days cycles: Pembrolizumab 200 mg IV day 1 of 21-day cycles
  In the event of PSA rise (25% increase over cycle 9 day 1, minimum of 2 ng/ml), and no evidence of radiographic progression, participants will receive 4 additional vaccine booster cycles: 100 µg pTVG-AR i.d days 1, 8 + 200 mg pembrolizumab IV day 1 of q 21-day cycles, for cycles 1 and 2 followed by 100 µg pTVG-HP i.d. days 1, 8 + 200 mg pembrolizumab IV day 1 in 21-day cycles, for cycles 3 and 4
  pTVG-HP: pTVG-HP is a plasmid DNA, produced in E. coli, that encodes the complementary deoxyribonucleic acid (cDNA) for human prostatic acid phosphatase (PAP).
  pTVG-AR: pTVG-AR is a plasmid DNA
  Pembrolizumab: Pembrolizumab is a human programmed death receptor-1 (PD-1)-blocking antibody indicated for the treatment of patients with multiple different types of cancer.
Period: Overall Study
Arm/Group | Arm 1: One DNA Vaccine | Arm 2: Two DNA Vaccines
Started | 30 | 30
Analysis Population | 30 | 30
Completed | 21 | 17
Not Completed | 9 | 13
Not completed — participants still on study | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: One DNA Vaccine | Arm 2: Two DNA Vaccines | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (9.5) | 72.4 (7.0) | 71.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The expected 6-months PFS rate in Arm 1 (pTVG-HP DNA vaccine and Pembrolizumab) in this participant population is 20-30%. It is hypothesized that adding pTVG-AR DNA vaccine (Arm 2) will increase the 6-months PFS rate to at least 55%.
  The 6-month PFS rate will be calculated for each study arm along with the corresponding two-sided 95% confidence interval which will be constructed using the Wilson score method. Participants who withdraw from the study without a progression or death event before the 6-month assessment will be excluded from this analysis. The stratified (by randomization strata) Mantel-Haenszel test will be used to compare the 6-months PFS rates between study arms.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: One DNA Vaccine | Arm 2: Two DNA Vaccines
Number analyzed (Participants) | 30 | 30
percentage of participants | 51 [30 to 69] | 45 [22 to 66]

2. Secondary Outcome: Overall Objective Response Rate
Description: The number of responses will be summarized in tabular format, stratified by study arm. Of note, objective response rate using radiographic criteria will apply only to subjects with RECIST measurable disease (i.e. not subjects with bone-only metastatic disease). Response rates will be calculated for each study arm along with the corresponding two-sided 95% confidence interval which will be constructed using the Wilson score method. The stratified (by randomization strata) Mantel-Haenszel test will be used to compare the overall objective response rates between study arms
Time Frame: up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: The number of responses will be summarized in tabular format, stratified by study arm. PSA Response Rates will be calculated for each study arm along with the corresponding two-sided 95% confidence interval which will be constructed using the Wilson score method.
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Secondary Outcome: Median Radiographic Progression-Free Survival
Description: Progression-Free Survival will be analyzed using the Kaplan-Meier method. Median PFS will be calculated for each study arm and reported along with the corresponding 95% confidence intervals will which will constructed using the nonparametric Brookmeyer and Crowley method. The stratified (by randomization strata) log-rank test will be used to compare PFS between study arms.
Time Frame: up to 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Median Duration of PSA and Objective Response
Description: Duration of PSA and objective response will be analyzed using the Kaplan-Maier method. The median duration of PSA and objective response will be calculated and report along with the corresponding 95% confidence interval which will be constructed using the nonparametric Brookmeyer-Crowley method.
Time Frame: up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival will be analyzed using the Kaplan-Meier method. OS will be calculated for each study arm and reported along with the corresponding 95% confidence intervals will which will constructed using the nonparametric Brookmeyer and Crowley method. The stratified (by randomization strata) log-rank test will be used to compare OS between study arms.
Time Frame: up to 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Antigen-Specific Th1 Immune Response
Description: The number and frequencies of antigen-specific Th1 immune responses will be summarized in tabular format for each study arm and both study arms combined. A generalized linear model with a logit link function will be used to evaluate whether antigen-specific Th1 immunity elicited with treatment to either antigen (PAP or AR) is associated with PSA response. The interaction term between treatment arm and antigen-specific Th1 immune will be included in this model.
Time Frame: up to 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Safety and Tolerability: Toxicity Rates
Description: Participants will be evaluated at each visit by a review of systems based on the most recent version of the NCI common toxicity criteria. Toxicities will be summarized by type and severity in tabular format. Toxicity rates (grade 2, grade 3, grade 4, grade ≥ 2, grade ≥ 3, etc.) will be calculated for each study arm and reported along the corresponding 95% confidence intervals. The 95% confidence intervals will be constructed using the Wilson score method. Fisher's exact test wi be used to compare toxicity rates between study arms.
Time Frame: up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: participants will be followed for up to 5 years
Description: All adverse events (including grade 1 events) with a frequency greater than 5 percent, and any adverse events with grade greater than grade 1, that were believed to be at least possibly related to treatment, are shown for patients treated in Arms 1 and 2. The numbers represent the number of patients experiencing a particular event at any point during the treatment period.
Arm/Group | Arm 1: One DNA Vaccine | Arm 2: Two DNA Vaccines
All-Cause Mortality (participants affected / at risk) | 19/30 | 13/30
Serious Adverse Events (participants affected / at risk) | 4/30 | 4/30
Other Adverse Events (participants affected / at risk) | 22/30 | 22/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: One DNA Vaccine (N=30) | Arm 2: Two DNA Vaccines (N=30)
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Cord Compression Event (Nervous system disorders) | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: One DNA Vaccine (N=30) | Arm 2: Two DNA Vaccines (N=30)
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Hyper or Hypothyroidism (Endocrine disorders) | 4 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 5
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
GE reflux (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
LFT changes/hepatitis (Gastrointestinal disorders) | 1 | 4
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Hyperglycemia (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 2 | 3
Fatigue (General disorders) | 6 | 13
Fever (General disorders) | 2 | 2
Injection Site Reaction (General disorders) | 4 | 2
Insomnia (General disorders) | 0 | 1
Pain (General disorders) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
CPK Increase (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 1
Horner's Syndrome (Nervous system disorders) | 0 | 1
Peripheral neuropathy (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04090528/Prot_SAP_000.pdf